CLINICAL TRIAL: NCT01368874
Title: Evaluation of the Ulthera® System for Lifting and Tightening the Face and Neck
Brief Title: Lifting and Tightening of the Face and Neck Utilizing the Ulthera® System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-110
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2014-04

CONDITIONS: Facial and Neck Skin Laxity
MeSH Terms: conditions — Facies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Ulthera® System treatment of the submental and submandibular regions at two treatment depths, and the lower neck region at one treatment depth.
  Interventions: Device: Ulthera® System treatment
- Group B (Active Comparator): Ulthera® System treatment of skin above the jawline, as well as the submental, submandibular and lower neck regions.
  Interventions: Device: Ulthera® System treatment
- Group C (Active Comparator): Ulthera® System treatment of the submental, submandibular, and the lower neck regions at two treatment depths.
  Interventions: Device: Ulthera® System treatment

INTERVENTIONS:
Device: Ulthera® System treatment — Single treatment of focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy

SUMMARY:
This prospective, multi-center, single treatment clinical trial evaluates the clinical outcomes associated with a non-invasive treatment to obtain lift and tightening of facial and neck tissue utilizing the Ulthera® System to deliver ultrasound energy in a focused manner below the surface of the skin.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to demonstrate the effectiveness of the Ulthera® System to obtain improvement in overall lifting and tightening of skin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years.
* Subject in good health.
* Skin laxity in the lower face and neck.
* Willingness and ability to comply with protocol requirements and return for follow-up visits.
* Provides written informed consent and HIPAA authorization.

Exclusion Criteria:

* Pregnant or lactating.
* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the face and lower neck.
* Excessive skin laxity on the face and neck.
* Significant scarring in areas to be treated.
* Significant open facial wounds or lesions.
* Severe or cystic acne on the face.
* Presence of a metal stent or implant in the facial area to be treated.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Baumann, M.D., Principal Investigator — Baumann Cosmetic and Research Institute; Brian Zelickson, M.D., Principal Investigator — Zel Skin and Laser Specialist
Locations (2):
- United States (2):
  - Baumann Cosmetic and Research Institute, Miami Beach, Florida
  - Zel Skin and Laser Specialists, Edina, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at two private medical clinics. Seventy-one 71 subjects enrolled, of which 64 subjects received study treatment February and July of 2011.
Pre-assignment Details: Seven enrolled subjects did not receive a complete study treatment. Six subjects were deemed screen failures, and one subject withdrew consent after receiving only a partial treatment. Sixty-four 64)subjects were assigned in a non-randomized fashion to each treatment group at the discretion of the PI.
Groups:
- Group A: Dual depth treatment on the submental and submandibular regions and single-depth treatment to the lower neck region
- Group B: Dual depth treatment of the platysmal muscle above the jawline, as well as dual depth treatment on the submental, submandibular and lower neck regions.
- Group C: Dual depth treatment on the submental, submandibular and lower neck regions.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 34 | 5 | 25
Completed | 31 | 5 | 24
Not Completed | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 34 | 5 | 25 | 64
Age, Continuous [Mean (Full Range); unit: years] | 55.06 (NA) [43 to 65] | 57.4 [49 to 62] | 55.2 [39 to 65] | 55.3 [39 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 5 | 24 | 61
  Male | 2 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 5 | 7
  Not Hispanic or Latino | 32 | 5 | 20 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Fitzpatrick Skin Type Score [Number; unit: Participants] — Skin Type I = White;very fair,red or blonde hair blue eyes;freckles;Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes;Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  Participants
    Type I | 6 | 0 | 4 | 10
    Type II | 18 | 5 | 8 | 31
    Type III | 10 | 0 | 12 | 22
    Type IV | 0 | 0 | 0 | 0
    Type V | 0 | 0 | 1 | 1
BMI [Mean (Full Range); unit: Kg/m^2] | 25.53 [19.04 to 32.76] | 22.49 [19.58 to 27.1] | 26.32 [18.47 to 36.44] | 25.60 [18.47 to 36.44]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Overall Lifting and Tightening of the Jowls and/or Neck Laxity
Description: Improvement in overall lifting and tightening of skin as determined by masked, qualitative assessment of photographs at 90 days post-treatment compared to baseline. Efficacy was based on the number of treated subjects assessed as improved in skin laxity, horizontal neck folds, neck sagging, texture and/or ptosis.
Time Frame: 90 Days post-treatment
Measure: Number; unit: participants
Groups:
- All Subjects Treated: Sixty-one (61) of 64 treated participants completed the 90-day study visit; 2 participants (1 each from Groups A and C)were lost-to-follow-up, 1 participant(Group A) missed the visit.
- Group A: Participants that received dual depth Ultherapy® treatment on the submental and submandibular regions, and single-depth treatment to the lower neck region. Thirty-two (32) of 34 Group A participants completed the 90-day study visit; two participants were lost-to-follow-up.
- Group B: Participants that received dual depth Ultherapy® treatment on the lower face, submental, submandibular, and lower neck regions.
- Group C: Participants that received dual depth Ultherapy® treatment on the submental, submandibular and lower neck regions. Twenty-four (24) of 25 participants completed the 90-day study visit; 1 participant was lost-to-follow-up
- Groups B/C: Combined participants from Groups B and C that received dual depth Ultherapy® treatment over all regions treated, i.e., platysmal muscle above the jawline, and submental, submandibular and lower neck regions.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 61 | 32 | 5 | 24 | 29
participants | 22 | 10 | 1 | 11 | 12

2. Secondary Outcome: Improvement in Overall Lifting and Tightening of Jowl and/or Neck Laxity, as Assessed by the Principal Investigator (PI) and the Subject Using the Global Aesthetic Improvement Scale, i.e., PGAIS and SGAIS, Respectively.
Description: At 60 days post-treatment, a PGAIS and SGAIS were completed based on a live assessment of the subject and a photographic assessment comparing post-treatment photos to baseline photos, to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse "Any Improvement" includes participants assessed in categories 1-3
Time Frame: 60 days post-treatment
Population: At 60 days post-treatment, the PI and subject completed a Global Aesthetic Improvement Scale (PGAIS and SGAIS, respectively)for comparison to pre-treatment.
Measure: Number; unit: percentage of participants improved
Groups:
- All Subjects Treated: Sixty-one (61) of 64 treated participants completed the 60- visit.
- Group A: Participants that received dual depth Ultherapy®® treatment on the submental and submandibular regions, and single-depth treatment to the lower neck region. Thirty-one (31) participants completed the 60-day study visit.
- Group B: Participants that received dual depth Ultherapy® treatment on the lower face,submental, submandibular, and lower neck regions. Five participants completed the 60-day study visit.
- Group C: Participants that received dual depth Ultherapy® treatment on the submental, submandibular and lower neck regions. Twenty-five (25) participants completed the 60-day study visit.
- Groups B/C: Combined participants from Groups B and C that received dual depth Ultherapy® treatment over all regions treated, i.e., platysmal muscle above the jawline, and submental, submandibular and lower neck regions. Thirty (30) participants completed the 60-day study visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 61 | 31 | 5 | 25 | 30
percentage of participants improved
  PGAIS - Improved to Very Much Improved, 60-Day | 63.9 | 74.2 | 40 | 56 | 53.3
  SGAIS - Improved to Very Much Improved, 60-Day | 67.2 | 61.3 | 80 | 72 | 73.3

3. Secondary Outcome: Improvement in Overall Lifting and Tightening of Jowl and/or Neck Laxity, as Assessed by the Principal Investigator (PI) and the Subject Using the Global Aesthetic Improvement Scale, i.e., PGAIS and SGAIS, Respectively.
Description: At 90 days post-treatment, a PGAIS and SGAIS were completed based on a live assessment of the subject and a photographic assessment comparing post-treatment photos to baseline photos, to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse "Any Improvement" includes participants assessed in categories 1-3
Time Frame: 90 days post-treatment
Population: At 90 days post-treatment, the PI and subject completed a Global Aesthetic Improvement Scale (PGAIS and SGAIS, respectively)for comparison to pre-treatment.
Measure: Number; unit: percentage of participants improved
Groups:
- All Subjects Treated: Sixty-one (61) of 64 treated participants completed the 90-day study visit.
- Group A: Participants that received dual depth Ultherapy®® treatment on the submental and submandibular regions, and single-depth treatment to the lower neck region. Thirty-two (32) participants completed the 90-day study visit.
- Group B: Participants that received dual depth Ultherapy® treatment on the lower face,submental, submandibular, and lower neck regions. Five participants completed the 90-day study visit.
- Group C: Participants that received dual depth Ultherapy® treatment on the submental, submandibular and lower neck regions. Twenty-four(24) participants completed the 90-day study visit.
- Groups B/C: Combined participants from Groups B and C that received dual depth Ultherapy® treatment over all regions treated, i.e., platysmal muscle above the jawline, and submental, submandibular and lower neck regions. Twenty-nine (29) participants completed the 90-day study visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 61 | 32 | 2 | 24 | 29
percentage of participants improved
  PGAIS - Improved to Very Much Improved, 90-Day | 78.7 | 78.1 | 40 | 87.5 | 79.3
  SGAIS - Improved to Very Much Improved, 90-Day | 68.9 | 65.6 | 60 | 75 | 72.4

4. Primary Outcome: Improvement in Overall Lifting and Tightening of the Jowls and/or Neck Laxity - RE-ANALYZED GROUP
Description: Improvement in overall lifting and tightening of skin as determined by masked, qualitative assessment of photographs at 90 days post-treatment compared to baseline. Efficacy was based on the number of treated subjects assessed as improved in skin laxity, horizontal neck folds, neck sagging, texture and/or ptosis.
  A data set of 42 of the 61 participants were re-analyzed. Data were removed for 19 participants whose pre-treatment and/or post-treatment photos were of poor photo quality, i.e., poor lighting, poor focus, poor positioning, creating the potential for biasing the masked assessment results.
Time Frame: 90 Days post-treatment
Measure: Number; unit: participants
Groups:
- All Subjects Treated: A data set of 42 of the 61 participants were re-analyzed. Data were removed for 19 participants whose pre-treatment and/or post-treatment photos were of poor photo quality, i.e., poor lighting, poor focus, poor positioning, creating the potential for biasing the masked assessment results.
- Group A: Participants that received dual depth Ultherapy® treatment on the submental and submandibular regions, and single-depth treatment to the lower neck region.
- Group B: Participants that received dual depth Ultherapy® treatment on the lower face,submental,submandibular,and lower neck regions.
- Group C: Participants that received dual depth Ultherapy® treatment on the submental, submandibular and lower neck regions.
- Groups B/C: Combined participants from Groups B and C that received dual depth Ultherapy® treatment over all regions treated, i.e., platysmal muscle above the jawline, and submental, submandibular, and lower neck regions.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 42 | 16 | 5 | 21 | 26
participants | 22 | 10 | 1 | 11 | 12

5. Other Pre Specified Outcome: Subjects' Assessment of Pain
Description: Subjects' sensory response to the Ulthera treatment exposures were recorded for each anatomical region treated using a validated Numeric Rating Scale (0-10), with 0 representing no pain and 10 representing the worst pain possible.
Time Frame: During Ulthera treatment
Measure: Mean (Full Range); unit: units on a scale
Groups:
- All Subjects Treated: Sixty-four 64) treated participants' assessment of pain was completed during the Ulthera® treatment.
Arm/Group | All Subjects Treated | Group A | Group B | Group C
Number analyzed (Participants) | 64 | 34 | 5 | 25
units on a scale
  Submental | 4 [0 to 4] | 4 [0 to 7] | 5 [4 to 6] | 4 [1 to 6]
  Submandibular | 4 [1 to 8] | 4 [1 to 8] | 5 [4 to 7] | 4 [2 to 7]
  Lower Neck | 5 [1 to 8] | 5 [1 to 8] | 6 [5 to 6] | 5 [2 to 7]
  Lower Face | NA [NA to NA] — Only Group B subjects were treated on the lower face; Group B data already displayed. | NA [NA to NA] — Group A subjects were not treated on the lower face; only Group B subjects. | 4 [2 to 5] | NA [NA to NA] — Group C subjects were not treated on the lower face; only Group B subjects.

6. Secondary Outcome: Improvement in Overall Lifting and Tightening of Jowl and/or Neck Laxity , as Assessed by the Principal Investigator (PI) and the Subject Using the Global Aesthetic Improvement Scale, i.e., PGAIS and SGAIS, Respectively.
Description: At 180 days post-treatment, a PGAIS and SGAIS were completed based on a live assessment of the subject and a photographic assessment comparing post-treatment photos to baseline photos, to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) describing an overall assessment as follows:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse "Any Improvement" includes participants assessed in categories 1-3
Time Frame: 180 days post-treatment
Population: At 180 days post-treatment, the PI and subject completed a Global Aesthetic Improvement Scale (PGAIS and SGAIS, respectively)for comparison to pre-treatment.
Measure: Number; unit: percentage of participants improved
Groups:
- All Subjects Treated: Sixty(60) of 64 treated participants completed the 180-day study visit.
- Group A: Participants that received dual depth Ultherapy®® treatment on the submental and submandibular regions, and single-depth treatment to the lower neck region. Thirty-one (31) participants completed the 180-day study visit.
- Group B: Participants that received dual depth Ultherapy® treatment on the lower face,submental, submandibular, and lower neck regions. Five participants completed the study visit.
- Group C: Participants that received dual depth Ultherapy® treatment on the submental, submandibular and lower neck regions. Twenty-four (24) participants completed the 180-day study visit.
- Groups B/C: Combined participants from Groups B and C that received dual depth Ultherapy® treatment over all regions treated, i.e., platysmal muscle above the jawline, and submental, submandibular and lower neck regions. Twenty-nine (29) participants completed the 180-day study visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 60 | 31 | 5 | 24 | 29
percentage of participants improved
  PGAIS - Improved to Very Much Improved, 180-Day | 66.7 | 42 | 80 | 95.8 | 93.1
  SGAIS - Improved to Very Much Improved, 180-Day | 63.3 | 54.8 | 40 | 79.2 | 72.4

7. Secondary Outcome: Patient Satisfaction 90 Days Post-treatment
Description: Patient satisfaction was determined by scores on a patient satisfaction questionnaire (PSQ) completed at 90 days post-treatment. Subjects indicated on a PSQ whether they saw improvement in the areas treated, i.e., providing a Yes/No response, and how satisfied they were with their Ulthera treatment, i.e., Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Pre-treatment and Day 90 post-treatment photographs were available for viewing during the assessment. Subjects also had a mirror in hand for real time assessment, comparing pre-treatment and 90 day post-treatment photos. Proportions of subjects reporting Improvement, and Very Satisfied and Satisfied are included.
Time Frame: 90 Days post-treatment
Measure: Number; unit: Percentage of participants
Groups:
- Group C: Participants that received dual depth Ultherapy® treatment on the submental, submandibular and lower neck regions. Twenty-four (24) participants completed the 90-day study visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 61 | 32 | 5 | 24 | 29
Percentage of participants
  Improvement Noticed | 82 | 81.3 | 80 | 83.3 | 82.8
  Very Satisfied + Satisfied | 65.6 | 62.5 | 40 | 75 | 68.9

8. Secondary Outcome: Patient Satisfaction Questionnaire 180 Days Post-treatment
Description: Patient satisfaction was determined by scores on a patient satisfaction questionnaire (PSQ) completed at 180 days post-treatment. Subjects indicated on a PSQ whether they saw improvement in the ares treated, i.e., providing a Yes/No response, and how satisfied they were with their Ulthera treatment, i.e., Very Satisfied, Satisfied, Dissatisfied, Very Dissatisfied. Pre-treatment and Day 180 post-treatment photographs were available for viewing during the assessment. Subjects also had a mirror in hand for real time assessment, comparing pre-treatment and 180 day post-treatment photos. Proportions of subjects reporting Improvement, and Very Satisfied and Satisfied are included.
Time Frame: 180 days post-treatment
Measure: Number; unit: Percentage of participants
Groups:
- All Subjects Treated: Sixty (60) of 64 treated participants completed the 180-day study visit.
- Group B: Participants that received dual depth Ultherapy® treatment on the lower face,submental, submandibular, and lower neck regions. Five participants completed the 180-day study visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 60 | 31 | 5 | 24 | 29
Percentage of participants
  Participants Reporting Improvement Noticed | 71.7 | 67.7 | 40 | 83.3 | 83.3
  Participants Very Satisfied + Satisfied | 55 | 41.9 | 40 | 75 | 68.9

9. Secondary Outcome: L'Oreal Photographic Scale Baseline
Description: At baseline, the Principal Investigator (PI) assessed the subjects' horizontal neck folds, neck sagging, and texture and ptosis changes using the L'Oreal Photographic Scales. The L'Oreal scales include the following categories, with a higher grade denoting an increased severity in each category:
  * Horizontal neck folds (Grades 0-6)
  * Neck sagging (Grades 0-7);
  * Texture (Female grades 0-5; male grades 0-7);
  * Ptosis (Female grades 0-5; males grades 0-7).
Time Frame: Baseline
Measure: Mean (Full Range); unit: units on a scale
Groups:
- All Subjects Treated: Treated subjects completing a 60 day post-treatment visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 64 | 34 | 5 | 25 | 30
units on a scale
  Horizontal Neck Folds | 3.0 [2 to 5] | 3.0 [2 to 5] | 3.8 [3 to 5] | 2.9 [2 to 4] | 3.1 [2 to 5]
  Neck Sagging | 3.7 [2 to 5] | 3.5 [2 to 5] | 4.2 [4 to 5] | 3.8 [3 to 5] | 3.9 [3 to 5]
  Texture | 2.8 [1 to 5] | 2.4 [1 to 5] | 3.2 [2 to 4] | 3.1 [2 to 5] | 3.1 [2 to 5]
  Ptosis | 3.2 [1 to 5] | 3.2 [1 to 5] | 3.6 [3 to 5] | 3.2 [2 to 5] | 3.3 [2 to 5]

10. Secondary Outcome: L'Oreal Photographic Scale 90 Days Post-treatment
Description: At 90 days post-treatment, the Principal Investigator (PI) assessed the subjects' horizontal neck folds, neck sagging, and texture and ptosis changes using the L'Oreal Photographic Scales. The L'Oreal scales include the following categories, with a higher grade denoting an increased severity in each category:
  * Horizontal neck folds (Grades 0-6)
  * Neck sagging (Grades 0-7);
  * Texture (Female grades 0-5; male grades 0-7);
  * Ptosis (Female grades 0-5; males grades 0-7).
Time Frame: 90 Days post-treatment
Measure: Mean (Full Range); unit: units on a scale
Groups:
- All Subjects Treated: Treated subjects completing a 90 day post-treatment visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 61 | 31 | 5 | 25 | 30
units on a scale
  Horizontal Neck Folds | 2.1 [1 to 5] | 2.6 [1 to 5] | 2.4 [2 to 3] | 1.5 [1 to 3] | 1.6 [1 to 3]
  Neck Sagging | 2.7 [0 to 6] | 3.0 [0 to 5] | 2.6 [1 to 4] | 2.4 [1 to 6] | 2.4 [1 to 6]
  Texture | 2.4 [1 to 5] | 2.3 [1 to 5] | 2.4 [2 to 4] | 2.6 [1 to 5] | 2.6 [1 to 5]
  Ptosis | 2.5 [0 to 5] | 2.8 [0 to 5] | 2.6 [1 to 3] | 2.1 [0 to 4] | 2.2 [0 to 4]

11. Secondary Outcome: L'Oreal Photographic Scale 180 Days Post-treatment
Description: At 180 days post-treatment, the Principal Investigator (PI) assessed the subjects' horizontal neck folds, neck sagging, and texture and ptosis changes using the L'Oreal Photographic Scales. The L'Oreal scales include the following categories, with a higher grade denoting an increased severity in each category:
  * Horizontal neck folds (Grades 0-6)
  * Neck sagging (Grades 0-7);
  * Texture (Female grades 0-5; male grades 0-7);
  * Ptosis (Female grades 0-5; males grades 0-7).
Time Frame: 180 Days post-treatment
Measure: Mean (Full Range); unit: units on a scale
Groups:
- All Subjects Treated: Treated subjects completing a 180 day post-treatment visit.
Arm/Group | All Subjects Treated | Group A | Group B | Group C | Groups B/C
Number analyzed (Participants) | 60 | 31 | 5 | 24 | 29
units on a scale
  Horizontal Neck Folds | 2.3 [0 to 5] | 2.7 [0 to 5] | 2.0 [1 to 3] | 1.7 [0 to 3] | 1.7 [0 to 3]
  Neck Sagging | 2.7 [0 to 5] | 3.2 [0 to 5] | 2.0 [1 to 3] | 2.2 [0 to 5] | 2.2 [0 to 5]
  Texture | 2.5 [1 to 5] | 2.3 [1 to 5] | 2.6 [1 to 4] | 2.6 [1 to 4] | 2.6 [1 to 4]
  Ptosis | 2.6 [1 to 5] | 3.0 [1 to 5] | 2.2 [1 to 3] | 2.2 [1 to 3] | 2.1 [1 to 4]

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C | Groups B/C
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/5 | 0/25 | 0/30
Other Adverse Events (participants affected / at risk) | 0/34 | 0/5 | 0/25 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less